CLINICAL TRIAL: NCT02880345
Title: RADVAX™: A Pilot Trial of Combined Pembrolizumab and Hypofractionated Radiation in Patients With Advanced Urothelial Cancer Who Have Progressed on Anti-PD-1/PD-L1 Monotherapy
Brief Title: RADVAX™: A Trial of Combined Pembrolizumab and Hypofractionated Radiation in Patients With Advanced Urothelial Cancer Who Have Progressed on Anti-PD-1/PD-L1 Monotherapy
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Insufficient accrual
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 22816
Record Dates: First submitted 2016-08-19; First posted 2016-08-26 (Estimated); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Urothelial Cancer
MeSH Terms: interventions — pembrolizumab; Radiation Dose Hypofractionation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 1 - 8 Gy x 3 fractions (Active Comparator): 8 Gy x 3 fractions
  Interventions: Drug: PEMBROLIZUMAB; Radiation: hypofractionated radiation
- Cohort 2 - 17 Gy x 1 fractions (Active Comparator): 17 Gy x 1 fraction
  Interventions: Drug: PEMBROLIZUMAB; Radiation: hypofractionated radiation

INTERVENTIONS:
Drug: PEMBROLIZUMAB
Radiation: hypofractionated radiation

SUMMARY:
This is a pilot study of a fixed dose of Pembrolizumab in combination with two different regimens of hypofractionated radiation. It is designed to demonstrate the activity and safety of the combination treatment in advanced urothelial cancer patients with prior exposure to PD-1 inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent/assent for the trial.
* Be 18 years of age or older on day of signing informed consent.
* Histologically confirmed diagnosis of pure or mixed urothelial cancer.
* Stage IV cancer by AJCC staging criteria. Patients who are stage IV as a result of cT4b disease only are not eligible.
* Progression of disease (radiographic or clinical) while on anti-PD-1 or anti-PD-L1 therapy at least 9 weeks or more from the date of starting anti-PD-1 or anti-PD-L1 therapy.
* Presence of an index lesion greater than or equal to 1 cm amenable to hypofractionated radiotherapy
* Patients who have metastatic cancer must have at least one lesion that is outside the radiation field that measures greater than one cm that can be followed by RECIST 1.1. This lesion, if it is close to the radiated lesion, must receive no more than 10% of the dose prescribed to the target lesion.
* Have provided tissue from an archival tissue sample or newly obtained core or excisional biopsy of a tumor lesion.
* Have a performance status of 0 or 1 on the ECOG Performance Scale.
* Ability to tolerate hypofractionated radiation therapy (e.g. lie flat and hold position)
* Demonstrate adequate organ function, all screening labs should be performed within 14 days of treatment initiation.
* Patients on dialysis are excluded from this study.
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for more than 1 year. 14. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria

* Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment. Systemic steroids administered specifically as a premedication for chemotherapy infusion or radiotherapy are allowed.
* Has had a prior monoclonal antibody within 4 weeks prior to study Day 1 or who has not recovered (i.e., less than or at Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., less than or at Grade 1 or at baseline) from adverse events due to a previously administered agent. - Note: Subjects with less than or Grade 2 neuropathy are an exception to this criterion and may qualify for the study. - Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* A history of prior radiotherapy that precludes delivery of hypofractionated radiotherapy
* Has a known additional malignancy that is progressing or requires active treatment.

Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.

* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment.
* Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjogrens syndrome will not be excluded from the study.
* Has evidence of interstitial lung disease or active, non-infectious pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subjects participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the prescreening or screening visit through 120 days after the last dose of trial treatment.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has received a live vaccine within 30 days prior to the first dose of trial treatment.
* Had progression of disease within 9 weeks of starting prior anti-PD-1 or anti-PD-L1 monotherapy therapy.
* Has not had prior cisplatinum-based chemotherapy, unless the subject is considered cisplatinum-ineligible based on meeting at least one of the following criteria: a. ECOG performance status of 2 (the proportion of ECOG 2 subjects will be limited to approximately 50% of the total population) b. Creatinine clearance (calculated or measured) less than 60 mL/min but greater than 30 mL/min Note: Subjects with a creatinine clearance (calculated or measured) less than 30 mL/min or on dialysis are excluded from the trial. c. CTCAE v.4, Greater than Grade 2 audiometric hearing loss (25dB in two consecutive wave ranges) d. CTCAE v.4, Greater than Grade 2 peripheral neuropathy e. NYHA Class III heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: John Christodouleous, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States